CLINICAL TRIAL: NCT01229176
Title: A Phase 2a, Randomized, Controlled, Observer Blind, Age De-Escalation, Multicenter and Multinational Study of the Safety, Reactogenicity and Immunogenicity of the NVGH Glycoconjugate Vaccine Against S. Typhi in Adults, Children, Older Infants and Infants
Brief Title: Safety and Immunogenicity of Vi-CRM197 Vaccine Against S. Typhi in Adults, Children, Older Infants and Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H01_02TP
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Typhoid Fever
MeSH Terms: conditions — Typhoid Fever | interventions — Polysaccharides; Vaccines; Pneumococcal Vaccines; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Vi-CRM, Adults (Experimental): Adults (18 to 45 years) receiving 1 dose of NVGH Vi-CRM197 vaccine
  Interventions: Biological: Vi-CRM197 vaccine
- Vi-PS, Adults (Active Comparator): Adults (18 to 45 years) receiving 1 dose of licensed Vi Polysaccharide vaccine
  Interventions: Biological: Vi Polysaccharide (PS) vaccine
- Vi-CRM, Children (Experimental): Children (24 to 59 months) receiving 2 doses of NVGH Vi-CRM197 vaccine
  Interventions: Biological: Vi-CRM197 vaccine
- Vi-PS, Children (Active Comparator): Children (24 to 59 months) receiving 1 dose of licensed Vi Polysaccharide vaccine and 1 dose of Pneumococcal conjugate vaccine
  Interventions: Biological: Vi Polysaccharide (PS) vaccine; Biological: Pneumococcal conjugate vaccine
- Vi-CRM, Older infants (Experimental): Older Infants (9 to 12 months) receiving 2 doses of NVGH Vi-CRM197 vaccine
  Interventions: Biological: Vi-CRM197 vaccine
- PNC13, Older infants (Active Comparator): Older Infants (9 to 12 months) receiving 2 doses of Pneumococcal conjugate vaccine
  Interventions: Biological: Pneumococcal conjugate vaccine
- Vi-CRM, Infants (Experimental): Infants (6 to 8 weeks) receiving 3 doses of NVGH Vi-CRM197 vaccine
  Interventions: Biological: Vi-CRM197 vaccine
- PNC13, Infants (Active Comparator): Infants (6 to 8 weeks) receiving 3 doses of Pneumococcal conjugate vaccine
  Interventions: Biological: Pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: Vi-CRM197 vaccine
  Arms: Vi-CRM, Adults; Vi-CRM, Children; Vi-CRM, Infants; Vi-CRM, Older infants
Biological: Vi Polysaccharide (PS) vaccine
  Other Names: Typherix
  Arms: Vi-PS, Adults; Vi-PS, Children
Biological: Pneumococcal conjugate vaccine
  Other Names: Prevenar 13
  Arms: PNC13, Infants; PNC13, Older infants; Vi-PS, Children

SUMMARY:
This phase 2 trial is aimed to obtain information on the safety and immunogenicity of the Vi-CRM197 in subjects from various age groups in India and Pakistan where Typhoid Fever is highly endemic and an efficacious vaccine against this disease is very much needed.

ELIGIBILITY:
Main eligibility criteria:

* Subjects belonging to 4 age groups will be enrolled into the trial: adults (18 to 45 years of age), children (24 to 59 months of age), older infants (9 to 12 months of age at enrollment) and infants (6 weeks of age at enrolment).
* Written informed consent will be obtained by the all subjects or their parents/ guardians (depending on the age group) before enrollment into the trial.
* Only females with a negative pregnancy test and willing to participate in family planning consultations (organized by the site study team) will be allowed to participate to the trial.
* Infants who have been vaccinated with 1 dose of BCG, HBV and OPV at birth can be enrolled into the trial, while infants who have received DTwP+HBV+Hib or OPV due at 6 weeks of age as per local EPI schedule cannot be enrolled into the trial.

Ages: 6 Weeks to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NVGH, Study Director — Novartis
Locations (2):
- K.E.M. Hospital Research Centre, Pune, Maharashtra, India
- The Aga Khan University Hospital, Karachi, Pakistan

REFERENCES:
- [Result] Bhutta ZA, Capeding MR, Bavdekar A, Marchetti E, Ariff S, Soofi SB, Anemona A, Habib MA, Alberto E, Juvekar S, Khan RM, Marhaba R, Ali N, Malubay N, Kawade A, Saul A, Martin LB, Podda A. Immunogenicity and safety of the Vi-CRM197 conjugate vaccine against typhoid fever in adults, children, and infants in south and southeast Asia: results from two randomised, observer-blind, age de-escalation, phase 2 trials. Lancet Infect Dis. 2014 Feb;14(2):119-29. doi: 10.1016/S1473-3099(13)70241-X. Epub 2013 Nov 28. PMID 24290843

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vi-CRM, Adults | Vi-PS, Adults | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Started | 40 | 40 | 20 | 20 | 20 | 20 | 20 | 20
Completed | 40 | 37 | 20 | 19 | 18 | 18 | 20 | 17
Not Completed | 0 | 3 | 0 | 1 | 2 | 2 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Vi-CRM, Adults | Vi-PS, Adults | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants | Total
Number analyzed (Participants) | 40 | 40 | 20 | 20 | 20 | 20 | 20 | 20 | 200
Age, Customized [Number; unit: participants]
  6 weeks to 8 weeks (infants) | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20 | 40
  9 months to 12 months (older infants) | 0 | 0 | 0 | 0 | 20 | 20 | 0 | 0 | 40
  24 months 59 months (children) | 0 | 0 | 20 | 20 | 0 | 0 | 0 | 0 | 40
  18 years to 45 years (adults) | 40 | 40 | 0 | 0 | 0 | 0 | 0 | 0 | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 11 | 9 | 12 | 12 | 10 | 8 | 97
  Male | 22 | 23 | 9 | 11 | 8 | 8 | 10 | 12 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 40 | 40 | 20 | 20 | 20 | 20 | 20 | 20 | 200
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Pakistan | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 160
  India | 20 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least 4-fold Increase in Anti-Vi Enzyme-linked Immunosorbent Assay (ELISA) Titer
Time Frame: At 28 days after last vaccination as compared to baseline
Population: Intention-to-treat analysis set, which included all participants who received the vaccination, those in whom at least one post-vaccination blood sample was collected, and those for whom at least one ELISA result was available.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Vi-CRM, Adults | Vi-PS, Adults | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Number analyzed (Participants) | 40 | 40 | 19 | 19 | 20 | 17 | 20 | 17
percentage of subjects | 100 [91 to 100] | 85 [70 to 94] | 100 [82 to 100] | 89 [67 to 99] | 95 [75 to 100] | 0 [0 to 20] | 85 [62 to 97] | 6 [0 to 29]

2. Primary Outcome: Percentage of Subjects With at Least 4-fold Increase in Anti-Vi ELISA Titer
Time Frame: At 6 months after last vaccination as compared to baseline
Population: Intention-to-treat analysis set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Vi-CRM, Adults | Vi-PS, Adults | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Number analyzed (Participants) | 40 | 37 | 20 | 19 | 18 | 18 | 20 | 17
percentage of subjects | 90 [76 to 97] | 81 [65 to 92] | 95 [75 to 100] | 68 [43 to 87] | 89 [65 to 99] | 6 [0 to 27] | 25 [9 to 49] | 0 [0 to 20]

3. Primary Outcome: Anti-Vi ELISA Geometric Mean Concentration (GMC)
Time Frame: At 28 days after last vaccination
Population: Intention-to-treat analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units/mL
Arm/Group | Vi-CRM, Adults | Vi-PS, Adults | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Number analyzed (Participants) | 40 | 40 | 19 | 19 | 20 | 17 | 20 | 17
ELISA Units/mL | 153 [105 to 224] | 44 [30 to 65] | 136 [91 to 202] | 53 [36 to 79] | 109 [80 to 148] | 1.43 [1.03 to 2] | 23 [17 to 32] | 2.33 [1.63 to 3.32]

4. Primary Outcome: Anti-Vi ELISA GMC
Time Frame: At 6 months after last vaccination
Population: Intention-to-treat analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units/mL
Arm/Group | Vi-CRM, Adults | Vi-PS, Adults | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Number analyzed (Participants) | 40 | 37 | 20 | 19 | 18 | 18 | 20 | 17
ELISA Units/mL | 59 [40 to 87] | 36 [24 to 53] | 23 [15 to 34] | 25 [17 to 38] | 22 [14 to 33] | 3.12 [2.08 to 4.68] | 3.76 [2.77 to 5.08] | 1.41 [1.02 to 1.96]

5. Secondary Outcome: Number of Participants With Any Solicited Local and Systemic Reaction, After Any Vaccination
Description: Solicited local reactions were: Adults, children, older infants, infants: erythema, induration and pain/tenderness at the injection site.
  Solicited systemic reactions were: Adults: chills, malaise, myalgia, arthralgia, headache, fatigue, rash and fever.
  Children, older infants and infants: lethargy, irritability, vomiting, diarrhoea, loss of appetite, rash and fever (and persistent crying in infants).
Time Frame: During the 7-day follow-up period after vaccination
Population: Analysis was done on as treated safety population.
Measure: Number; unit: participants
Arm/Group | Vi-CRM, Adults | Vi-PS, Adults | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Number analyzed (Participants) | 40 | 40 | 20 | 20 | 20 | 20 | 20 | 19
participants | 24 | 27 | 18 | 17 | 14 | 19 | 20 | 19

ADVERSE EVENTS:
Time Frame: Solicited Adverse Events (AEs) were collected during 7-day follow period after each vaccination. Serious AEs were collected throughout the study period. Unsolicited AEs were collected collected during 28-day follow period after each vaccination.
Description: Analysis was done on as treated safety population
Arm/Group | Vi-CRM, Adults | Vi-PS, Adults | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 2/20 | 1/20 | 4/20 | 5/20 | 5/20 | 3/19
Other Adverse Events (participants affected / at risk) | 24/40 | 29/40 | 19/20 | 17/20 | 18/20 | 20/20 | 20/20 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vi-CRM, Adults (N=40) | Vi-PS, Adults (N=40) | Vi-CRM, Children (N=20) | Vi-PS, Children (N=20) | Vi-CRM, Older Infants (N=20) | PNC13, Older Infants (N=20) | Vi-CRM, Infants (N=20) | PNC13, Infants (N=19)
Pneumonia (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 1 | 2 | 5 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Febrile Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — systemic assessment for children, older infants and infants
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0
Measles (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vi-CRM, Adults (N=40) | Vi-PS, Adults (N=40) | Vi-CRM, Children (N=20) | Vi-PS, Children (N=20) | Vi-CRM, Older Infants (N=20) | PNC13, Older Infants (N=20) | Vi-CRM, Infants (N=20) | PNC13, Infants (N=19)
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0
Eye Pian (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pian (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 8
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 6 | 4 | 9 | 12 | 7 | 6 — systemic assessment for children, older infants and infants
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 4 | 2 | 3 — systemic assessment for children, older infants and infants
Chills (General disorders) | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 0 — systemic assessment for adults
Crying (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 — systemic assessment for older infants and infants
Fatigue (General disorders) | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 0 — systemic assessment for adults
Injection Site Erythema (General disorders) | 4 | 4 | 2 | 1 | 2 | 3 | 9 | 5
Injection Site Induration (General disorders) | 4 | 5 | 4 | 2 | 2 | 5 | 9 | 9
Injection Site Pain (General disorders) | 17 | 17 | 16 | 14 | 5 | 9 | 17 | 15
Irritability (General disorders) | 0 | 0 | 2 | 3 | 3 | 1 | 11 | 8 — systemic assessment for children, older infants and infants
Malaise (General disorders) | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 — systemic assessment for adults
Pyrexia (General disorders) | 1 | 1 | 7 | 3 | 9 | 7 | 11 | 5
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Eye Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 5 | 1 | 12 | 14 | 12 | 11
Measles (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Oral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 — systemic assessment for adults
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0 — systemic assessment for adults
Headache (Nervous system disorders) | 13 | 14 | 1 | 0 | 0 | 0 | 0 | 0 — systemic assessment for adults
Somnolence (Nervous system disorders) | 0 | 0 | 6 | 4 | 4 | 3 | 7 | 4 — systemic assessment for children, older infants and infants
Eating Disorder (Psychiatric disorders) | 0 | 0 | 4 | 2 | 3 | 2 | 6 | 5 — systemic assessment for children, older infants and infants
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 6 | 3 | 8 | 8 | 10 | 6
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 12
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Heat Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 4 | 2 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event that no publication of the Study results has been made by NVGH within twelve (12) months of Study database lock and no proposed publication is under discussion by the publication committee, Principal Investigator may publish its own Study results.